CLINICAL TRIAL: NCT06421233
Title: The Effect of Endorphin Massage Applied to Postpartum Women on Anxiety and Fatigue Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Nurseli Soylu Erener, Research Assistant, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2023/516
Record Dates: First submitted 2024-05-08; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Birth; Anxiety; Fatigue
Keywords: Birth; Vaginal Birth; Massage; anxiety; Endorphin; Fatigue
MeSH Terms: conditions — Anxiety Disorders; Fatigue | interventions — Massage

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): * Personal introduction form, state and trait anxiety scale and visual similarity scale for fatigue were applied.
  * Endorphin massage was applied twice by the researcher for 15 minutes every two hours.
  * After the endorphin massage applied for the second time, the visual similarity scale and the state and trait anxiety scale were applied again for fatigue.
  Interventions: Other: massage
- Control gruop (No Intervention): * A personal introduction form, state and trait anxiety scale, and visual similarity scale for fatigue were applied.
  * Two hours after the first evaluation, the visual similarity scale and the state and trait anxiety scale were applied again for fatigue.

INTERVENTIONS:
Other: massage — Endorphin massage will be given for 15 minutes every 2 hours.
  Other Names: endorphin massage
  Arms: Intervention group

SUMMARY:
The postpartum period, especially in the first few weeks, can be a difficult period for mothers to adapt to the new situation of having a baby. During this process, physiological, psychological and social changes occur in the mother's body. While many mothers adapt to these changes easily, some mothers may experience psychological disorders at different levels.Among these, anxiety and depression are the most common diseases. Anxiety can negatively affect mothers, especially during birth and the postpartum period.During the postpartum period, nurses have the opportunity to improve maternal and infant health by recognizing and treating anxiety.Physical symptoms associated with postpartum anxiety include fatigue, irritability, difficulty concentrating, and sleep disturbances. However, during the vaginal birth process, mothers may feel tired in the early postpartum period, as the pregnant woman spends a lot of energy by staying hungry for a long time. When the literature was examined, it was determined that endorphin massage reduces back pain in pregnant women, reduces anxiety level in pregnant women, accelerates the involution process in the postpartum period, and has positive effects on postpartum depression.Similar to endorphin massage, it has been determined that back massage reduces back pain in the postpartum period and provides the mother with both physiological and psychological relief. In addition, no study has been found examining the effect of endorphin massage applied to postpartum women on anxiety levels and fatigue in the postpartum period. Therefore, this study aimed to determine the effect of endorphin massage applied to postpartum women who gave birth vaginally on postpartum anxiety and fatigue levels.

DETAILED DESCRIPTION:
Birth is a very important experience in a woman's life. The postpartum period is a period of 6-8 weeks after birth. During this process, physiological, psychological and social changes occur in the puerperal woman's body. While many postpartum women easily adapt to these changes, some postpartum women may experience psychological disorders at different levels. Anxiety can negatively affect postpartum women, especially during birth and the postpartum period. Although it is generally desirable to experience anxiety at a normal and mild level, excessive anxiety can tire the individual emotionally.In addition, postpartum women may feel tired in the early postpartum period due to the pregnant woman fasting for a long time and spending too much energy during the vaginal birth process.This situation can be caused by many physical, psychological and situational factors. Postpartum fatigue can lead to deterioration in the general health of the mother and her baby, as well as other serious problems.Postpartum fatigue negatively affects women's physical and mental functions, wound healing, self-care skills and behaviors, energy, motivation and cognitive status, adaptation to motherhood, baby care behaviors, relationships with marriage and family members, including sexuality, work performance and quality of life. is a symptom.In this process, applications applied to postpartum women increase the quality of life by reducing fatigue.Endorphin massage is among the practices performed to improve the quality of life of women during the postpartum period. Endorphin is a natural painkiller known as the happiness hormone, which is similar to opioids secreted by the body, reduces pain, provides relaxation, protects the body against infections, accelerates metabolism. It is known that massage increases endorphin levels by having a relaxing effect on the muscles. Endorphin massage increases the release of endorphins, allowing the individual to relax, relaxing the muscles and reducing pain. Endorphin massage is a light massage technique that can increase the release of oxytocin and endorphin hormones and provide a feeling of calmness and comfort. When the literature was examined, it was determined that endorphin massage reduces back pain in pregnant women, reduces anxiety level in pregnant women, accelerates the involution process in the postpartum period, and has positive effects on postpartum depression.Similar to endorphin massage, it has been determined that back massage reduces back pain in the postpartum period and provides the mother with both physiological and psychological relief. In addition, no study has been found examining the effect of endorphin massage applied to postpartum women on anxiety levels and fatigue in the postpartum period. Therefore, this study aimed to determine the effect of endorphin massage applied to postpartum women who gave birth vaginally on postpartum anxiety and fatigue levels.

ELIGIBILITY:
Inclusion Criteria:

* Giving birth vaginally at term,
* Postpartum within 24 hours,
* Primiparous,
* Those who are healthy and have given birth to a single baby,
* Postpartum women who volunteered to participate in the study were included.

Exclusion Criteria:

* Those with psychiatric illness (Bipolar Disorder, Depression, Obsessive Compulsive Disorder),
* People with chronic diseases (Heart disease, Thyroid problems, Diabetes mellitus, Hypertension, asthma, COPD,
* Those who have been diagnosed with a risky pregnancy (Pre-eclampsia, Arthritis, Pregnancy-related hypertension, Gestational diabetes),
* Whose baby was admitted to neonatal intensive care,
* Postpartum women with postpartum bleeding were not included in the study.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-09-04 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
State and Trait Anxiety Scale | It was applied twice in total, two hours apart.
  The state anxiety scale determines how the individual feels at a certain moment and under certain conditions. The scale consists of 20 questions and is asked to choose one of the options 'not at all', 'somewhat', 'a lot' and 'completely' depending on the severity of the thoughts or behaviors. The trait anxiety scale determines how the individual feels, regardless of the situation and conditions, and consists of 20 questions. In answering this scale, one is asked to choose one of the following options: 'almost never', 'sometimes', 'most of the time' and 'almost always', depending on the frequency of the thoughts or behaviors.

SECONDARY OUTCOMES:
Visual Similarity Scale for Fatigue | It was applied twice in total, two hours apart.
  The scale has sub-dimensions of fatigue and energy . It consists of a total of 18 items in two sub-dimensions.
  The scale consists of 10 cm horizontal lines with positive expressions at one end and negative expressions at the other end of each item. While the items of the fatigue sub-dimension progress from positive to negative expressions, the items of the energy sub-dimension are in the opposite order. The lowest score obtained in the fatigue sub-dimension is zero and the highest score is 130. In the energy sub-dimension, scores are calculated between 0 and 50 points. A high score of the fatigue sub-dimension and a low score of the energy sub-dimension indicate that the severity of fatigue increases.

CONTACTS AND LOCATIONS:
Overall Officials: Nurseli SOYLU ERENER, Principal Investigator — TC Erciyes University
Locations (1):
- Kayseri City Hospital, Kocasinan, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Only the name of the research can be shared.

REFERENCES:
- See also: Qian, J., Sun, S., Liu, L., & Yu, X. (2021). Protocol: Effectiveness of non-pharmacological interventions for reducing postpartum fatigue: a systematic review protocol. BMJ Open, 11(10), 51136 — http://doi.org/10.1136/BMJOPEN-2021-051136